CLINICAL TRIAL: NCT06650982
Title: The Effects of PechaKucha Presentation About Medical Device-Related Pressure Injuries on Knowledge and Attitudes of Nursing Students: a Randomized Controlled Study
Brief Title: The Effects of PechaKucha Presentation About Medical Device-Related Pressure Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MAİDE YEŞİLYURT (Other)
Responsible Party: Sponsor-Investigator, MAİDE YEŞİLYURT, DOCTOR, Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: MYESİLYURT4
Record Dates: First submitted 2024-05-15; First posted 2024-10-21 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Medical Device Site Injury
Keywords: pecha kucha; medical device related pressure injury; nursing student

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental arm (Experimental): Before medical device related pressure injury (MDRPI) training is given to students, an introductory characteristics form and knowledge and attitude surveys will be applied (pre-test). The survey questions will be administered immediately after the PK training presentation containing MDRPI information is given to the students (Posttest 1), and 4 weeks later (Posttest 2).
  Interventions: Other: Pecha Kucha presentation on MDPRI
- control arm (No Intervention): Before students are given MDRPI training, an introductory characteristics form and knowledge and attitude surveys will be administered (pre-test). The survey questions will be administered immediately after the traditional educational presentation containing MDRPI information is given to the students (Posttest 1), and again 4 weeks later (Posttest 2).

INTERVENTIONS:
Other: Pecha Kucha presentation on MDPRI — Students in the experimental arm will be given training on MDRPI.
  Other Names: EDUCATION RELATED TO MDRPI
  Arms: experimental arm

SUMMARY:
In the literature, no research has been found examining the knowledge and attitudes of students regarding medical device related pressure injury education given using the PK method. In addition to contributing to the existing literature, this research will also contribute to determining the effect of TAIBY training given with PK, a current presentation technique, on the learning and attitude levels of nursing students.

DETAILED DESCRIPTION:
Medical device-associated pressure injuries occur on the tissue and mucous membranes due to the pressure created by the medical device, but differ from other pressure injuries in that they do not occur on bone protrusions. European Pressure Injury Advisory Panel (EPUAP), The National Pressure Injury Advisory Panel (NPIAP) and the Pan Pacific Pressure Injury Alliance (PPPIA) define these injuries as "pressure injuries caused by tools used for diagnosis or treatment." It can develop in any anatomical region it comes into contact with, especially the ear, foot, neck, head and face. It is known that medical device-related pressure injuries constitute approximately one-third of the pressure injuries in hospitalized adult patients. Prevention and care interventions in medical device-related pressure injuries should be carried out in line with proven recommendations. is important for patient safety.

pread Pecha kucha (PK) is an innovative form of presentation used around the world (Byrne, 2016). PK, derived from the Japanese word meaning "chat", helps present creative works with visual images Pecha kucha is a compact and effective presentation method consisting of 20 slides, each presented in 20 seconds This "20×20" format, which requires careful editing and develops the use of critical communication skills, serves as an innovative and valuable tool that allows the presenter to dynamically and systematically present important information worth sharing to the audience . Thanks to Pecha Kucha, the presenter conveys the topic quickly and clearly without deviating from the essence of the topic Beyer et al. (2012) reported that PK may be superior to traditional PowerPoint presentations in terms of learning function. Klentzin et al. (2010) also stated that PK is as effective as traditional PowerPoint presentations in retaining information. It is stated that with the pecha kucha method, information can be presented in a more concise way, without any difference in quality, compared to a longer PowerPoint presentation

. PK presentation, including visual and narrative presentation, does not take more than 7-8 minutes It is stated that the use of the PK method is effective in transferring theoretical content into practice and providing emotional learning in nursing education (Byrne, 2016). Students studying in health services were given training on the prevention of pressure injuries with the PK presentation method, and it was determined that the knowledge level of the students increased with the PK method . In a study comparing PK and traditional presentation in nursing education, it was found that there was no difference between the two methods, but it was recommended that the PK method be used on issues that require attention In studies using PK in medical education, it was stated that the majority of students liked this learning method and wanted it to be used in other courses .

In the literature, no research has been found examining the knowledge and attitudes of students regarding medical device related pressure ınury education given using the PK method. In addition to contributing to the existing literature, this research will also contribute to determining the effect of training given with PK, a current presentation technique, on the learning and attitude levels of nursing students.

ELIGIBILITY:
Inclusion Criteria:

* Being a nursing student
* volunteer

Exclusion Criteria:

* Not being a nursing student
* not volunteering

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-11-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Pressure injury knowledge level of students | up to 4 weeks
  students' "Medical Device-related Pressure Sore Knowledge Level Assessment Test score",
students' pressure injury attitude level | up to 4 weeks
  students' "Pressure Injury Attitude Survey Regarding Medical Devices score"

CONTACTS AND LOCATIONS:
Overall Officials: Serpil YUKSEL, PHD, Study Chair — Necmettin Erbakan University
Locations (1):
- Aksaray University, Merkez, Turkey (Türkiye)